CLINICAL TRIAL: NCT00305110
Title: Safety and Speed of Onset of a Fixed Dose of Intravenous Hydromorphone in the Treatment of Adult Patients Presenting to the Emergency Department With Acute Severe Pain
Brief Title: Safety of Hydromorphone in Adult Patients Presenting to the Emergency Department With Acute Severe Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Chang, MD, MD, Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMC 0511307; NCT01006850 (obsolete NCT alias)
Record Dates: First submitted 2006-03-17; First posted 2006-03-21 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Acute Pain
Keywords: Pain; Acute; Emergency Department; Severe; Hydromorphone; Dilaudid; Adult
MeSH Terms: conditions — Acute Pain; Pain; Emergencies; Lymphoma, Follicular | interventions — Hydromorphone

ARMS (1):
- 2 mg IV hydromorphone (Experimental): 2 mg IV hydromorphone administered over 2-3 minutes
  Interventions: Drug: 2 mg IV hydromorphone

INTERVENTIONS:
Drug: 2 mg IV hydromorphone
  Other Names: Dilaudid

SUMMARY:
The purpose of this study is to determine the safety and speed of onset of 2mg intravenous hydromorphone (Dilaudid) in patients weighing at least 150 lbs presenting to the emergency department with acute severe pain

DETAILED DESCRIPTION:
Introduction and Background: Pain is cited as the most frequent reason for visits to emergency departments (EDs) (McCaig, 2001). It can be estimated from the National Hospital Ambulatory Medical Care Survey, an annual survey of a representative sample of visits to US EDs, that there are 17 million visits per year to US EDs for specific complaints of pain, 29 million visits including "back symptoms" and "injuries not otherwise specified" as well as specific mentions of pain. However it is widely acknowledged that pain is seriously under-treated in the ED as well as in other health care settings (Ducharme, 1996; Selbst, 1990; Wilson, 1989). The concern regarding under-treatment is reflected in new standards for pain management developed by the Joint Commission on Accreditation of Healthcare Organizations (JCAHO) requiring assessment of pain at triage in the ED and referring to pain measurement as the "fifth vital sign" (Philips, 2000).

Proper pain management is a tremendous challenge to ED physicians as pain is not only a noxious experience but also a symptom of injury and disease that needs to be understood and appropriately treated. Further complicating pain management is the large interpersonal variability in pain perception and expression reflecting cultural, contextual, and individual differences between people. Reasons for under-treating pain include concern over side effects of opioids, perception of pain complaints as possible drug-seeking behavior, under-staffing, concern that analgesics will mask symptoms or delay early diagnosis and treatment, and contribute to risks of tolerance and dependence in vulnerable patients.

Morphine has long been considered the gold standard in pain control. Hydromorphone is another powerful opioid that has been used extensively for the management of post-operative pain and morphine-resistant cancer-related pain. A recent Cochrane review on the use of hydromorphone found 32 studies that focused on acute pain (Quigley, 2003). Of these 32 studies, only 9 involved intravenous forms of hydromorphone (Coda, 1997; Collins, 1996; Deutsch, 1968; Jasani, 1994; Liu, 1995; Mahler, 1975; Rapp, 1996; Searle, 1994; Urquhart, 1988). Of these 8 studies, 5 involved patient controlled analgesia, and only 1 study compared IV hydromorphone to IV morphine (Mahler, 1975). The Cochrane review concludes that there are substantial gaps in the understanding of the efficacy and potency of hydromorphone.

We have recently completed a study in non-elderly adult patients (IRB 04-08-225) that showed that weight-based IV hydromorphone provides better pain relief than weight-based IV morphine. This result was both statistically and clinically significant. We also demonstrated in this same study that IV hydromorphone has a faster onset and also provided statistically significant improvement in pain relief at 5 minutes as compared to IV morphine.

Although weight-based dosing of medications is common in pediatrics, most emergency physicians use whole integer amounts of pain medications. IV hydromorphone is more potent than IV morphine, so the dosages given are much smaller. We therefore wish to give a standard 2 mg dose of IV hydromorphone to all non-elderly adult patients weighing at least 150 lbs presenting to the ED with acute severe pain. We wish to examine the safety and speed of onset of hydromorphone using such a protocol.

Our general thought is that to develop more evidence based practice, we need to generate more practice based evidence. This study attempts to do this as it is practiced based and very practical. We wish to take the drug as it comes (2mg Dilaudid in an ampule) and use all of it, thus alleviating the need to waste the excess opioid (and alleviating the need to find a second person to witness the wasting). We also wish to use a weight cutoff that everyone can remember (150 lbs). We believe that this protocol will provide greater pain relief and help address the issue of inadequate pain treatment, or "oligoanalgesia", that is prominent in the literature (Sobel 2002, Wilson, 1989, Goldfrank 2000).

Finally, in our multiple studies of pain conducted in the ED, we have found a relatively high rate of refusal to receive pain medication. We think this may represent a component to the problem of oligoanalgesia that is widespread in the ED. We wish to investigate the reasons for patient refusal to receiving parental opioid medications (fear of addiction, side effects, etc).

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 21 years
2. Age less than 65 years of age
3. Pain with onset within 7 days
4. ED attending physician's judgment that patient's pain warrants use of morphine
5. Normal mental status

Exclusion Criteria:

1. Prior use of methadone
2. Use of other opioids or tramadol within past seven days
3. Prior adverse reaction to hydromorphone.
4. Chronic pain syndrome
5. Alcohol intoxication
6. SBP <90 mm Hg
7. Use of MAO inhibitors in past 30 days
8. C02 measurement greater than 46

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2006-01; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew K Chang, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 2 mg IV Hydromorphone: 2 mg IV hydromorphone administered over 2-3 minutes
  2 mg IV hydromorphone
Period: Overall Study
Arm/Group | 2 mg IV Hydromorphone
Started | 298
All Necessary Data Collected | 269
Completed | 269
Not Completed | 29
Not completed — Missing data | 29

BASELINE CHARACTERISTICS:
Population: 29 participants had missing data and were excluded from analysis
Arm/Group | 2 mg IV Hydromorphone
Number analyzed (Participants) | 269
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166
  Male | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 163
  African-American | 85
  White | 16
  Other | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 269
Pain Location [Count of Participants; unit: Participants]
  Abdomen | 205
  Other | 64
Baseline Pain intensity [Count of Participants; unit: Participants] — Pain intensity is measured on a numerical rating scale (NRS) from 0 (no pain) to 10 (worst pain imaginable).
  Participants
    less than 7 | 10
    7 | 22
    8 | 45
    9 | 33
    10 | 158
Weight [Mean (Standard Deviation); unit: pounds] | 198 (38)
Final diagnosis [Count of Participants; unit: Participants]
  Abcess | 7
  Appendicitis | 18
  Biliary colic/cholecystitis | 21
  Diverticulitis | 14
  Gastritis | 8
  Kidney Stone | 38
  Low back pain | 7
  Nonspecific abdominal pain | 65
  Pancreatitis | 9
  Pyelonephritis | 6
  Small bowel obstruction | 8
  Other | 68
Disposition [Count of Participants; unit: Participants] — Disposition is where the participant goes after the ED. Discharge means they are well enough to leave the hospital. Admit means they were admitted to the hospital for an inpatient stay. Against medical advice means that although the physician recommended they come into the hospital for an inpatient stay, the patient chose to leave the hospital and go against the recommendation of their doctor.
  Participants
    Admitted | 122
    Discharged | 144
    Against medical advice | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Requiring Naloxone
Description: Naloxone is a reversal agent - a medication that reverses the effects of another. Hydromorphone is an opiate pain medication that acts as a depressant to the body, thereby slowing it down. A large slow down is dangerous, as it can cause the breathing rate to slow down too much and prevent enough oxygen from entering the body and reaching the brain, resulting in death. Naloxone is a medication that blocks the receptors binding opiate pain medication and reversing the body's reaction to the hydromorphone, allowing body processes to return to normal speeds, including the breathing rate. The use of naloxone in the study indicates that the participant received too much pain medication or reacted more strongly than the average person, requiring the rescue medication to reverse the negative effects. The number of participants who required naloxone is assessed.
Time Frame: immediately after infusion, up to 120 minutes post infusion
Measure: Count of Participants; unit: Participants
Arm/Group | 2 mg IV Hydromorphone
Number analyzed (Participants) | 269
Participants | 0

2. Secondary Outcome: Number of Participants Experiencing a Respiratory Rate Lower Than 12 Breaths Per Minute
Description: Normal respiratory rate ranges from 12 to 20 breaths per minute. The decreased respiration results in a decreased amount of oxygen entering the body and therefore low amount of oxygen supplied to the brain. Prolonged oxygen deprivation can result in injury or death. Respiratory rates lower than 12 breaths per minute is a sign of distress. Number of participants experiencing a respiratory rate lower than 12 breaths per minute is measured.
Time Frame: immediately after infusion, up to 120 minutes post infusion
Measure: Count of Participants; unit: Participants
Arm/Group | 2 mg IV Hydromorphone
Number analyzed (Participants) | 269
Participants | 12

3. Secondary Outcome: Number of Participants Experiencing a Systolic Blood Pressure Less Than 90 mmHg
Description: Normal systolic blood pressure is approximately 120 mmHg. A low systolic blood pressure indicates blood, and therefore oxygen, are not being distributed around the body properly. This leads to a decreased amount of oxygen for the body to use and can result in injury or death if prolonged or severe.
Time Frame: Immediately after infusion, up to 120 minutes post infusion
Measure: Count of Participants; unit: Participants
Arm/Group | 2 mg IV Hydromorphone
Number analyzed (Participants) | 269
Participants | 2

4. Secondary Outcome: Oxygen Desaturation Measured Over 2-hour Time Frame
Description: blood oxygen saturation less than 95% is considered oxygen desaturation. Blood oxygen saturation is normally above 95%. Oxygen desaturation of less than 90% is dangerous because there is less oxygen throughout the body for cellular energy. Prolonged or severe blood oxygen desaturation can result in injury or death.
Time Frame: immediately after infusion, up to 120 minutes post infusion
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | 2 mg IV Hydromorphone
Number analyzed (Participants) | 296
participants
  at least 95% oxygen saturation, all time points | 68 [62 to 73]
  90-94% oxygen saturation, one or more times | 26 [21 to 32]
  below 90% oxygen saturation, one or more times | 6 [4 to 10]

5. Secondary Outcome: Oxygen Saturation Measured Over 2-hour Time Frame
Description: blood oxygen saturation is measured periodically from 1 minute to 120 minutes after the medication was infused
Time Frame: baseline to 120 minutes post infusion
Measure: Median (Inter-Quartile Range); unit: % oxygen saturation
Arm/Group | 2 mg IV Hydromorphone
Number analyzed (Participants) | 269
% oxygen saturation
  Baseline | 99 [98 to 100]
  1 minute post infusion | 98 [96 to 99]
  2 minutes post infusion | 98 [96 to 99]
  3 minutes post infusion | 98 [96 to 99]
  4 minutes post infusion | 98 [96 to 99]
  5 minutes post infusion | 97 [96 to 99]
  15 minutes post infusion | 97 [96 to 99]
  30 minutes post infusion | 98 [96 to 99]
  120 minutes post infusion | 98 [97 to 99]

6. Post Hoc Outcome: Pain Intensity Assessed Over 2-hour Time Frame
Description: Pain intensity is measured on the numerical rating scale (NRS), from 0 ("no pain") to 10 ("worst pain possible"). Participants are asked to rate their pain periodically over a 2 hour time period following infusion of the medication.
Time Frame: baseline up to 120 minutes after post infusion
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | 2 mg IV Hydromorphone
Number analyzed (Participants) | 269
units on a scale
  Baseline | 10 [8 to 10]
  1 minute post infusion | 4 [0 to 7]
  2 minutes post infusion | 3 [0 to 6]
  3 minutes post infustion | 3 [0 to 5]
  4 minutes post infusion | 2 [0 to 5]
  5 minutes post infusion | 1 [0 to 5]
  15 minutes post infusion | 1 [0 to 4]
  30 minutes post infusion | 0 [0 to 3]
  120 minutes post infusion | 1 [0 to 4]

ADVERSE EVENTS:
Time Frame: 120 minutes
Arm/Group | 2 mg IV Hydromorphone
All-Cause Mortality (participants affected / at risk) | 0/269
Serious Adverse Events (participants affected / at risk) | 0/269
Other Adverse Events (participants affected / at risk) | 100/269
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 2 mg IV Hydromorphone (N=269)
Respiratory Rate <12 breathes per minute (Respiratory, thoracic and mediastinal disorders) | 12
Heart Rate <60 beats/min (Vascular disorders) | 34
Systolic blood pressure <90 mmHg (Vascular disorders) | 2
Nausea (Gastrointestinal disorders) | 21/125 — excluding patients who were nauseated or had vomited at baseline, before receiving hydromorphone
Vomiting (Gastrointestinal disorders) | 9/125 — excluding patients who were nauseated or had vomited at baseline, before receiving hydromorphone
Pruritis (Skin and subcutaneous tissue disorders) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes